CLINICAL TRIAL: NCT06300827
Title: The Effect of Structured Digital-Based Education Given to Nursing Students on Disaster Literacy and Disaster Preparedness Belief Level: A Randomized Controlled Trial
Brief Title: The Effect of Structured Digital-Based Education Given to Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Naile Bilgili, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023 - 1302
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: 18 Years and Over

STUDY DESIGN:
Intervention Model Description: Experimental Group: Structured digital-based training will be implemented. Control Group: The nursing student will be expected to continue their daily life.
  Nursing students who meet the inclusion criteria will be randomly assigned to the experimental group by a statistician.
Who Masked: Outcomes Assessor
Masking Description: Research data/output measurements are made by a research assistant not involved in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group: Structured digital-based training will be implemented.
  Interventions: Other: Structured digital-based training
- Control Group (No Intervention): Control Group: The nursing student will be expected to continue their daily life.
  Nursing students who meet the inclusion criteria will be randomly assigned to the experimental group by a statistician.

INTERVENTIONS:
Other: Structured digital-based training — The eight week intervention will be delivered in 15 different sessions, each session lasting 40 minutes. It is expected that the seventh week session will last approximately 150 minutes. The control group is expected to continue with their daily lives.
  Arms: Experimental Group

SUMMARY:
Turkey is a risky country in terms of disasters. Preparedness and awareness for all disasters affecting the whole world gain value. Disaster literacy is an important approach to evaluating disaster preparedness and awareness processes. Disaster literacy is defined as the ability of an individual to access, read, understand, and use the information necessary to make informed decisions and follow instructions in the context of mitigation, preparation, response, and recovery during a disaster Disaster literacy needs to be increased to raise awareness among individuals and minimize disaster risk. Along with the awareness studies, it is also important to identify the disaster preparedness belief in order to encourage individuals to change potentially harmful behavior. Belief in disaster preparedness; It may vary according to the perception of experiencing a disaster, the perceived severity of the disaster, the benefits of being prepared for a disaster, the perceived barriers to being prepared for a disaster, being prepared, and the individual's belief in his or her ability to cope with a disaster. It may be useful to determine both disaster preparedness beliefs and disaster literacy levels of individuals at the social level. It is predicted that when multiple interventions are brought together in the learning process, there will be a faster and more lasting effect. In this study, which aims to use education and information technology together, a structured digital-based educational intervention is planned. The intervention program was structured by taking advantage of both the advantages of the digital world and active learning methods in order to keep the student active. The program is eight weeks and consists of seven dimensions and the purpose of the program is based on accessing information, understanding, information, making decisions, and applying information. The planned study aimed to determine the effect of structured digital-based education given to university students studying in the nursing department on their disaster literacy and disaster preparedness belief levels.

DETAILED DESCRIPTION:
Study protocol Nursing students who meet the inclusion criteria will be pre-tested and post-tested. The first test will be administered at baseline and the last test will be administered at week 8. The eight-week intervention will be delivered in 15 different sessions, each session lasting 40 minutes. It is expected that the seventh-week session will last approximately 150 minutes. The control group is expected to continue with their daily lives. There will be no intervention by the researcher during the research process. After the research is completed, the research team will hold an information meeting with the control group about the structured digital-based training content, and the materials used in the research will be given to the control group. The study will use simple randomization. https://www.random.org/ will be used to allocate students who meet the inclusion criteria to a specified number of groups. The data/outcome measures of the study (evaluator) will be blinded in terms of statisticians and reporting. Data collection tools: Personal Information Form, Disaster Literacy Scale, General Disaster Preparedness Belief Levels Scale based on the Health Belief Model.

ELIGIBILITY:
Inclusion criteria

* To be enrolled in the nursing programme
* Ability to speak and understand Turkish
* Speak English at least at beginner level
* To have signed the informed consent form

Exclusion criteria

* Having previously participated in any disaster training programme
* Failure to attend the eight-week digital-based disaster training programme twice in a row

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Disaster Literacy Scale | Baseline, Weeks 8
  It is a self-report scale designed to assess disaster literacy in people aged 18-60. The conceptual framework of the 61-item scale consists of 16 domains. Each item is scored 1-5 (1 - very difficult, 2 - difficult, 3 - undecided, 4 - easy, 5 - very easy). The total score that can be obtained from the scale is between 61 and 305. An increase in the score obtained from the scale means that the participant's level of disaster literacy is increasing. For ease of calculation, the total score is standardised to a value between 0-50. The scale is divided into metrics as 0-<30 points insufficient, 30-<36 points limited, 36-<42 points sufficient and 42-50 points excellent disaster literacy.
General Disaster Preparedness Belief Scale Using the Health Belief | Baseline, Weeks 8
  The purpose of the scale is to assess individuals' emergency/disaster preparedness behaviours, attitudes and beliefs based on the Health Belief Model. Individuals over the age of 18 can participate in the scale. The scale has a total of 31 items and 6 sub-dimensions. These sub-dimensions are 'perceived sensitivity', 'perceived seriousness', 'perceived benefits', 'perceived barriers', 'action motivators' and 'self-efficacy'. All items are rated on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). There are 14 negative items on the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bilgili, Study Director — Gazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Gazi University, Ankara
  - Necmettin Erbakan University, Konya
  - Tokat Gaziosmanpaşa University, Tokat Province

REFERENCES:
- [Derived] Genc FZ, Yildiz S, Erdal A, Bilgili N. Effect of structured digital-based education given to nursing students on disaster literacy and disaster preparedness belief levels: A randomized controlled study. Nurse Educ Today. 2025 Apr;147:106581. doi: 10.1016/j.nedt.2025.106581. Epub 2025 Jan 17. PMID 39837253